CLINICAL TRIAL: NCT04193709
Title: Effects of Activity-Dependent Plasticity on Recovery of Bladder and Sexual Function After Human Spinal Cord Injury
Brief Title: Recovery of Bladder and Sexual Function After Human Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Charles Hubscher, Professor, University of Louisville
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19.1194; OT2OD024898 (NIH)
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Urinary Bladder, Neurogenic; Blood Pressure; Autonomic Dysreflexia; Bowel Incontinence
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Autonomic Dysreflexia; Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: Cross-sectional and observational (Arm 1) Prospective, cohort, and interventional (Arm 2).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Measure symptomatic indices of autonomic dysreflexia (No Intervention): The purpose of this arm is to systematically measure symptomatic indices of autonomic nervous system activation and corresponding cardiovascular changes in persons with spinal cord injuries during bladder filling and bowel stimulation.
- Cardiovascular spinal cord epidural stimulation (Experimental): The purpose of this arm is to use spinal cord epidural stimulation for maintenance of blood pressure and heart rate in the lab during cystometry (bladder filling) and anorectal filling (bowel distension) and in the at-home setting for maintenance of normative blood pressure and heart rate that can be triggered from bladder filling and during bowel evacuation.
  Interventions: Device: Spinal Cord Epidural Stimulation

INTERVENTIONS:
Device: Spinal Cord Epidural Stimulation — For arm 2, optimal stimulation parameters (cathode/anode configuration, stimulation frequency and voltage; placement of electrode from L1 to S1) will be identified for blood pressure and bladder pressure to achieve a bladder capacity in the target normative range of 400-450 mLs. Spinal cord epidural stimulation will then be used in a controlled lab setting for the regulation of blood pressure and heart rate to maintain normative values (target systolic pressure of 110-120 mmHg) and bladder pressure below 10 cmH2O during bladder filling up to the targeted capacity (fill volume of 400 mLs).
  Arms: Cardiovascular spinal cord epidural stimulation

SUMMARY:
This study will incorporate critical cross viscero-visceral intersystem interactions to 1) investigate in a controlled laboratory setting and then with mobile at-home monitoring the extent, severity, and frequency of occurrence of autonomic dysreflexia with respect to daily bladder and bowel function, in conjunction with identifying potential underlying mechanisms by examining urinary biomarkers for several specific vasoactive hormones, and 2) to regulate cardiovascular function therapeutically as part of bladder and bowel management using spinal cord epidural stimulation.

ELIGIBILITY:
Arm 1 Inclusion Criteria:

* At least 18 years of age;
* AIS A to D;
* Neurogenic bladder and bowel dysfunction;
* Stable medical condition

Arm 2 Inclusion Criteria:

* At least 18 years of age;
* AIS A to D;
* Neurogenic bladder and bowel dysfunction;
* Use of intermittent catheterization for bladder emptying;
* Prior implantation of a Medtronic scES array

Arms 1 and 2 Exclusion Criteria:

* Prior Botox injections of the bladder and/or bladder augmentation surgery;
* Colostomy bag,
* Ventilator dependent;
* Any implanted pump (i.e. Baclofen pump, pain pump, etc.);
* Pregnant at the time of enrollment or planning to become pregnant during the time course of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2026-01-03 (Estimated); Study Completion 2027-01-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in systolic blood pressure over a 24 hour period after 80 sessions (6 months) | Baseline, 80 sessions (6 months)
  We will record systolic blood pressure every five minutes over a 24 hour period using a 24-hour blood pressure monitor

SECONDARY OUTCOMES:
Change from baseline in bladder capacity after 80 sessions (6 months) | Baseline, 80 sessions (6 months)
  Using urodynamics we will measure bladder capacity in mL
Change from baseline in detrusor pressure after 80 sessions (6 months) | Baseline, 80 sessions (6 months)
  Using urodynamics we will measure detrusor pressure in cmH2O.
Change from baseline in mean resting anal pressure after 80 sessions (6 months) | Baseline, 80 sessions (6 months)
  Using anorectal manometry will will measure mean resting anal pressure in mmHg.
Change from baseline in mean squeeze pressure after 80 sessions (6 months) | Baseline, 80 sessions (6 months)
  Using anorectal manometry we will measure mean squeeze pressure in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hubscher, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No